CLINICAL TRIAL: NCT03687684
Title: Randomized, Double-Blind, Placebo-Controlled, Phase 1 Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single and Multiple Doses of TAK 831 in Healthy Adult Asian Subjects
Brief Title: Phase 1 Study of TAK-831 in Healthy Adult Asian Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Other
Other Study IDs: TAK-831-1002; U1111-1219-2623 (Other: WHO); JapicCTI-184127 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2018-09-26; First posted 2018-09-27 (Actual); Results first posted 2020-06-29 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Japanese Cohort 1-A; TAK-831 100 mg + TAK-831 300 mg (Experimental): TAK-831 100 milligrams (mg), tablets, orally, once daily on Day 1, followed by TAK-831 300 mg, tablets, orally, once daily on Day 9 in healthy Japanese participants.
  Interventions: Drug: TAK-831
- Japanese Cohort 1-B; TAK-831 100 mg + Placebo (Experimental): TAK-831 100 mg, tablets, orally, once daily on Day 1 followed by TAK-831 matching placebo, tablets, orally, once daily on Day 9 in healthy Japanese participants.
  Interventions: Drug: TAK-831; Drug: Placebo
- Japanese Cohort 1-C; Placebo + TAK-831 300 mg (Experimental): TAK-831 matching placebo, tablets, orally, once daily on Day 1 followed by TAK-831 300 mg, tablets, orally, once daily on Day 9 in healthy Japanese participants.
  Interventions: Drug: TAK-831; Drug: Placebo
- Japanese Cohort 2; TAK-831 300 mg (Experimental): TAK-831 300 mg or TAK-831 matching placebo, tablets, orally, once daily on Day 1 followed by TAK-831 300 mg or TAK-831 matching placebo, tablets, orally, once daily from Day 4 to Day 17 in healthy Japanese participants.
  Interventions: Drug: TAK-831; Drug: Placebo
- Chinese Cohort 3; TAK-831 600 mg (Experimental): TAK-831 600 mg or TAK-831 matching placebo, tablets, orally, once daily on Day 1 followed by TAK-831 600 mg or TAK-831 matching placebo, tablets, orally, once daily from Day 4 to Day 17 in healthy Chinese participants. This cohort is optional and will be decided to run based on the data of Cohorts 1 and 2. The dose will be defined based on the result of Cohort 1 or Cohort 2.
  Interventions: Drug: TAK-831; Drug: Placebo
- Japanese Cohort 4; TAK-831 600 mg (Experimental): TAK-831 600 mg or TAK-831 matching placebo, tablets, orally, once daily on Day 1 followed by TAK-831 600 mg or TAK-831 matching placebo, tablets, orally, once daily from Day 4 to Day 17 in healthy Japanese participants. This cohort is optional and will be decided to run based on the data of Cohorts 1 and 2. The dose will be defined based on the result of Cohort 1 or Cohort 2.
  Interventions: Drug: TAK-831; Drug: Placebo
- Japanese Cohort 5; TAK-831 (Experimental): TAK-831 50 mg or TAK-831 matching placebo, tablets, orally, once daily on Day 1 followed by TAK-831 50 mg or TAK-831 matching placebo, tablets, orally, once daily from Day 4 to Day 17 in healthy Japanese participants.
  Interventions: Drug: TAK-831; Drug: Placebo

INTERVENTIONS:
Drug: TAK-831 — TAK-831 Tablets.
Drug: Placebo — TAK-831 Matching Placebo Tablets.
  Arms: Chinese Cohort 3; TAK-831 600 mg; Japanese Cohort 1-B; TAK-831 100 mg + Placebo; Japanese Cohort 1-C; Placebo + TAK-831 300 mg; Japanese Cohort 2; TAK-831 300 mg; Japanese Cohort 4; TAK-831 600 mg; Japanese Cohort 5; TAK-831

SUMMARY:
The purpose of this study is to evaluate safety, tolerability, pharmacokinetics, and pharmacodynamics of TAK-831 when administered as single or multiple oral doses in healthy adult Asian participants.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-831. This study will assess the safety, tolerability, pharmacokinetics (PK), and Pharmacodynamics (PD) of TAK-831 when administered as single or multiple oral doses in healthy adult Asian participants (Japanese and Chinese participants).

The study will enroll approximately 40 participants and include up to 5 cohorts of healthy adult Japanese or Chinese participants as following (8 participants per a cohort). Cohorts 3, 4 and 5 are optional and will be decided to run based on the data of Cohorts 1 and 2. Dose level for these cohorts will be defined based on the result of Cohort 1 or Cohort 2.

* Japanese Cohort 1-A; TAK-831 100 mg single dose + TAK-831 300 mg single dose
* Japanese Cohort 1-B; TAK-831 100 mg single dose + Placebo single dose
* Japanese Cohort 1-C; Placebo single dose + TAK-831 300 mg single dose
* Japanese Cohort 2; TAK-831 300 mg or TAK-831 matching placebo, single dose + TAK-831 300 mg or TAK-831 matching placebo, multiple dose *
* Chinese Cohort 3; TAK-831 600 mg or TAK-831 matching placebo, single dose + TAK-831 600 mg or TAK-831 matching placebo, multiple dose
* Japanese Cohort 4; TAK-831 600 mg or TAK-831 matching placebo, single dose + TAK-831 600 mg or TAK-831 matching placebo, multiple dose
* Japanese Cohort 5; TAK-831 50 mg or TAK-831 matching placebo, single dose + TAK-831 50 mg or TAK-831 matching placebo, multiple dose *The dose in Cohort 2 will be adjusted based on the safety and tolerability as well as PK and PD in Cohort 1.

Above all treatment, randomization information will remain undisclosed to the participant and study doctor during the study (unless there is an urgent medical need) and TAK-831 will be administered orally.

This single center trial will be conducted in Japan. The overall time to participate in Cohort 1 of this study is approximately 12 days and 19 days in Cohorts 2 to 5. 11 days (for Cohort 1) or 12 days (for Cohorts 2 to 5) after last dose of study drug, participants will be contacted by telephone for a follow-up assessment unless abnormal, clinically significant findings are observed upon discharge.

ELIGIBILITY:
Inclusion Criteria:

1. The participant must understand the study procedures and agree to participate by providing written informed consent (for Chinese participants, an interpreter should be present as necessary).
2. The participant must be willing and able to comply with all study procedures and restrictions.
3. The participant must be male or female (of nonchildbearing potential) aged 20 to 55 years, inclusive, at the Screening.
4. The participant must have a body mass index (BMI) >=18.5 kg/m^2 and =<25.0 kg/m^2 at the Screening.
5. The participant must be a current nonsmoker who has not used tobacco- or nicotine-containing products (e.g., nicotine patch) for at least 6 months prior to the Screening.
6. Chinese participants are defined as participants who were born in mainland China, and their biological parents and grandparents must all have been of Chinese origin (for Cohort 3 only).
7. Chinese participants who have lived out of China for more than 5 years must not have significantly modified their diets since leaving China (for Cohort 3 only).
8. The participant must be judged to be in good health by the investigator, based on clinical evaluations including laboratory tests, medical history, full physical examination, 12-lead electrocardiogram, and vital sign measurements performed at the Screening and prior to the first dose of study drug.
9. The participant must meet the birth control requirements.

Exclusion Criteria:

1. The participant has a history of clinically significant endocrine, gastrointestinal (including motility disorder and intestinal obstruction), cardiovascular, hematological, hepatic, immunological, renal, respiratory, or genitourinary, or presents with major neurological (including stroke and chronic seizures) abnormalities or diseases.
2. The participant has participated in another investigational trial within 4 weeks before the pretrial visit (Screening). The 4-week window will be derived from the date of the last trial procedure and/or adverse event (AE) related to the trial procedure in the previous trial to the Screening Visit of the current trial.
3. The participant is an employee or immediate family member (e.g., spouse, parent, child, sibling) of the sponsor.
4. The participant has a history of cancer (malignancy).
5. The participant has a history of significant multiple and/or severe allergies (e.g., food, drug, latex allergy) or has had an anaphylactic reaction or significant intolerability to prescription or nonprescription drugs or food.
6. The participant has a positive alcohol or drug or immunological screen.
7. The participant is of childbearing potential or lactating.
8. The participant had major surgery, received or lost 1 unit of blood (approximately 500 milliliters [mL]) within 8 weeks prior to the first dose of study drug.
9. The participant with any gastrointestinal (GI) surgery that could impact upon the absorption of study drug.
10. The participant has a known hypersensitivity to any component of the formulation of TAK-831 or related compounds.
11. The participant is unable to refrain from or anticipates the use of any medication, including prescription and nonprescription drugs or herbal remedies, beginning approximately 7 days before administration of the initial dose of trial drug, throughout the trial (including washout intervals between trial periods), until the Follow-up Visit.
12. The participant has a history of alcohol consumption exceeding 2 standard drinks per day on average (1 glass is approximately equivalent to: beer [354 mL/12 ounces], wine [118 mL/4 ounces], or distilled spirits [29.5 mL/1 ounce] per day).
13. The participant who consumes excessive amounts, defined as greater than 6 servings (1 serving is approximately equivalent to 120 mg of caffeine) of coffee, tea, cola, energy drinks, or other caffeinated beverages per day.
14. The participant has a history of drug abuse.
15. The participant has a (QT interval with Fridericia's correction method) QTcF >450 milliseconds (msec) (males) or >470 msec (females) or PR outside the range of 120 to 220 msec at the Screening Visit or Check-in.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-10-09 (Actual); Primary Completion 2019-06-09 (Actual); Study Completion 2019-06-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Hospital Tokyo, Shinjuku-ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at single site in Japan from 09 October 2018 to 19 June 2019.
Pre-assignment Details: Healthy adult participants were randomized to receive TAK-831: under 3-sequential dose escalation design to the sequence of administration of A (100 mg +300 mg), B (100 mg + Placebo), and C (Placebo + 300 mg) in Cohort 1 (Japanese); single dose followed by multiple dose of TAK-831 or Placebo in Cohorts 2, 4, 5 (Japanese) and in Cohort 3 (Chinese).
Groups:
- Japanese Cohort 1-A: TAK-831 100 mg + TAK-831 300 mg: TAK-831 100 milligram (mg), tablet, orally, once on Day 1 of Part 1, followed by TAK-831 300 mg, tablet, orally, once on Day 1 (Day 9) of Part 2 in healthy Japanese participants.
- Japanese Cohort 1-B: TAK-831 100 mg + Placebo: TAK-831 100 mg, tablet, orally, once on Day 1 of Part 1 followed by TAK-831 matching placebo, tablet, orally, once on Day 1 (Day 9) of Part 2 in healthy Japanese participants.
- Japanese Cohort 1-C: Placebo + TAK-831 300 mg: TAK-831 matching placebo, tablet, orally, once on Day 1 of Part 1 followed by TAK-831 300 mg, tablet, orally, once on Day 1 (Day 9) of Part 2 in healthy Japanese participants.
- Japanese Cohort 2, 4 and 5: Pooled Placebo: TAK-831 matching placebo, tablet, orally, once on Day 1 and once daily from Day 4 to Day 17 in healthy Japanese participants.
- Japanese Cohort 2: TAK-831 300 mg: TAK-831 300 mg, tablet, orally, once on Day 1 and once daily from Day 4 to Day 17 in healthy Japanese participants.
- Japanese Cohort 4: TAK-831 600 mg: TAK-831 600 mg, tablet, orally, once on Day 1 and once daily from Day 4 to Day 17 in healthy Japanese participants.
- Japanese Cohort 5: TAK-831 50 mg: TAK-831 50 mg, tablet, orally, once on Day 1 and once daily from Day 4 to Day 17 in healthy Japanese participants.
- Chinese Cohort 3: Placebo: TAK-831 matching placebo, tablet, orally, once on Day 1 and once daily from Day 4 to Day 17 in healthy Chinese participants.
- Chinese Cohort 3: TAK-831 600 mg: TAK-831 600 mg, tablet, orally, once on Day 1 and once daily from Day 4 to Day 17 in healthy Chinese participants.
Period: Overall Study
Arm/Group | Japanese Cohort 1-A: TAK-831 100 mg + TAK-831 300 mg | Japanese Cohort 1-B: TAK-831 100 mg + Placebo | Japanese Cohort 1-C: Placebo + TAK-831 300 mg | Japanese Cohort 2, 4 and 5: Pooled Placebo | Japanese Cohort 2: TAK-831 300 mg | Japanese Cohort 4: TAK-831 600 mg | Japanese Cohort 5: TAK-831 50 mg | Chinese Cohort 3: Placebo | Chinese Cohort 3: TAK-831 600 mg
Started | 4 | 2 | 2 | 6 | 6 | 6 | 6 | 2 | 6
Completed | 4 | 2 | 2 | 6 | 6 | 6 | 6 | 2 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set was defined as all participants who received at least one dose of study drug.
Groups:
- Japanese Cohort 1-A: TAK-831 100 mg + TAK-831 300 mg: TAK-831 100 mg, tablet, orally, once on Day 1 of Part 1, followed by TAK-831 300 mg, tablet, orally, once on Day 1 (Day 9) of Part 2 in healthy Japanese participants.
- Total: Total of all reporting groups
Arm/Group | Japanese Cohort 1-A: TAK-831 100 mg + TAK-831 300 mg | Japanese Cohort 1-B: TAK-831 100 mg + Placebo | Japanese Cohort 1-C: Placebo + TAK-831 300 mg | Japanese Cohort 2, 4 and 5: Pooled Placebo | Japanese Cohort 2: TAK-831 300 mg | Japanese Cohort 4: TAK-831 600 mg | Japanese Cohort 5: TAK-831 50 mg | Chinese Cohort 3: Placebo | Chinese Cohort 3: TAK-831 600 mg | Total
Number analyzed (Participants) | 4 | 2 | 2 | 6 | 6 | 6 | 6 | 2 | 6 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 2 | 2 | 6 | 6 | 6 | 6 | 2 | 6 | 40
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 4 | 2 | 2 | 6 | 6 | 6 | 6 | 2 | 6 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 4 | 2 | 2 | 6 | 6 | 6 | 6 | 2 | 6 | 40
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 4 | 2 | 2 | 6 | 6 | 6 | 6 | 2 | 6 | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting at Least One Treatment-emergent Adverse Event (TEAE)
Time Frame: Cohort 1: Baseline up to Day 23; Cohorts 2-5: Baseline up to Day 31
Population: The safety analysis set was defined as all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Japanese Cohort 1: Placebo: TAK-831 matching placebo, tablets, orally, once on Day 1 of Part 1 and Day 1 (Day 9) of Part 2 in healthy Japanese participants.
- Japanese Cohort 1: TAK-831 100 mg: TAK-831 100 mg, tablet, orally, once on Day 1 of Part 1 in healthy Japanese participants.
- Japanese Cohort 1: TAK-831 300 mg: TAK-831 300 mg, tablet, orally, once on Day 1 (Day 9) of Part 2 in healthy Japanese participants.
Arm/Group | Japanese Cohort 1: Placebo | Japanese Cohort 1: TAK-831 100 mg | Japanese Cohort 1: TAK-831 300 mg | Japanese Cohort 2, 4 and 5: Pooled Placebo | Japanese Cohort 2: TAK-831 300 mg | Japanese Cohort 4: TAK-831 600 mg | Japanese Cohort 5: TAK-831 50 mg | Chinese Cohort 3: Placebo | Chinese Cohort 3: TAK-831 600 mg
Number analyzed (Participants) | 4 | 6 | 6 | 6 | 6 | 6 | 6 | 2 | 6
Participants | 0 | 2 | 0 | 4 | 4 | 1 | 2 | 1 | 2

2. Primary Outcome: Number of Participants Reporting at Least One TEAE Related to Laboratory Test Results
Time Frame: Cohort 1: Baseline up to Day 23; Cohorts 2-5: Baseline up to Day 31
Population: The safety analysis set was defined as all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Japanese Cohort 1: Placebo | Japanese Cohort 1: TAK-831 100 mg | Japanese Cohort 1: TAK-831 300 mg | Japanese Cohort 2, 4 and 5: Pooled Placebo | Japanese Cohort 2: TAK-831 300 mg | Japanese Cohort 4: TAK-831 600 mg | Japanese Cohort 5: TAK-831 50 mg | Chinese Cohort 3: Placebo | Chinese Cohort 3: TAK-831 600 mg
Number analyzed (Participants) | 4 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 2
Participants | 0 | 2 | 0 | 2 | 2 | 1 | 1 | 1 | 0

3. Primary Outcome: Number of Participants Reporting at Least One TEAE Related to Vital Sign
Time Frame: Cohort 1: Baseline up to Day 23; Cohorts 2-5: Baseline up to Day 31
Population: The safety analysis set was defined as all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Japanese Cohort 1: Placebo | Japanese Cohort 1: TAK-831 100 mg | Japanese Cohort 1: TAK-831 300 mg | Japanese Cohort 2, 4 and 5: Pooled Placebo | Japanese Cohort 2: TAK-831 300 mg | Japanese Cohort 4: TAK-831 600 mg | Japanese Cohort 5: TAK-831 50 mg | Chinese Cohort 3: Placebo | Chinese Cohort 3: TAK-831 600 mg
Number analyzed (Participants) | 4 | 6 | 6 | 6 | 6 | 6 | 6 | 2 | 6
Participants | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants Reporting at Least One TEAE Related to Body Weight
Time Frame: Cohort 1: Baseline up to Day 23; Cohorts 2-5: Baseline up to Day 31
Population: The safety analysis set was defined as all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Japanese Cohort 1: Placebo | Japanese Cohort 1: TAK-831 100 mg | Japanese Cohort 1: TAK-831 300 mg | Japanese Cohort 2, 4 and 5: Pooled Placebo | Japanese Cohort 2: TAK-831 300 mg | Japanese Cohort 4: TAK-831 600 mg | Japanese Cohort 5: TAK-831 50 mg | Chinese Cohort 3: Placebo | Chinese Cohort 3: TAK-831 600 mg
Number analyzed (Participants) | 4 | 6 | 6 | 6 | 6 | 6 | 6 | 2 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants Reporting at Least One TEAE Related to 12-lead Electrocardiogram (ECG) Parameters
Time Frame: Cohort 1: Baseline up to Day 23; Cohorts 2-5: Baseline up to Day 31
Population: The safety analysis set was defined as all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Japanese Cohort 1: Placebo | Japanese Cohort 1: TAK-831 100 mg | Japanese Cohort 1: TAK-831 300 mg | Japanese Cohort 2, 4 and 5: Pooled Placebo | Japanese Cohort 2: TAK-831 300 mg | Japanese Cohort 4: TAK-831 600 mg | Japanese Cohort 5: TAK-831 50 mg | Chinese Cohort 3: Placebo | Chinese Cohort 3: TAK-831 600 mg
Number analyzed (Participants) | 4 | 6 | 6 | 6 | 6 | 6 | 6 | 2 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-831
Time Frame: Cohort 1: Day 1 pre-dose and at 0.5, 1, 1.5, 2, 4, 8, 12, 24, 36, 48 and 72 hours post-dose; Cohorts 2 to 5: Day 1 pre-dose and at 0.25, 0.5, 1, 1.5, 2, 4, 8, 12, 24, 36, 48 and 72 hours post-dose
Population: The pharmacokinetic (PK) analysis set included participants who received at least one dose of study drug, and who were appropriately evaluable for at least 1 PK parameter.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Japanese Cohort 1: TAK-831 100 mg | Japanese Cohort 1: TAK-831 300 mg | Japanese Cohort 2: TAK-831 300 mg | Japanese Cohort 4: TAK-831 600 mg | Japanese Cohort 5: TAK-831 50 mg | Chinese Cohort 3: TAK-831 600 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
nanogram per milliliter (ng/mL) | 985.5 (20.8) | 1823 (53.7) | 981.7 (29.1) | 1602 (42.1) | 339.9 (33.3) | 1807 (28.5)

7. Secondary Outcome: Cohorts 2 to 5, Cmax, ss: Maximum Observed Steady-state Plasma Concentration During a Dosing Interval for TAK-831
Time Frame: Day 17 pre-dose and at 0.25, 0.5, 1, 1.5, 2, 4, 8, 12 and 24 hours post-dose
Population: The PK analysis set included participants who received at least one dose of study drug, and who were appropriately evaluable for at least 1 PK parameter.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Japanese Cohort 2: TAK-831 300 mg | Japanese Cohort 4: TAK-831 600 mg | Japanese Cohort 5: TAK-831 50 mg | Chinese Cohort 3: TAK-831 600 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
ng/mL | 831.8 (29.1) | 1903 (33.6) | 417.0 (23.8) | 1581 (42.4)

8. Secondary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-831
Time Frame: Cohort 1: Day 1 pre-dose, 0.5, 1, 1.5, 2, 4, 8, 12, 24, 36, 48, 72 hours post-dose; Cohorts 2 to 5: Day 1 pre-dose, 0.25, 0.5, 1, 1.5, 2, 4, 8, 12, 24, 36, 48, 72 hours post-dose; Day 17 pre-dose, 0.25, 0.5, 1, 1.5, 2, 4, 8, 12, 24 hours post-dose
Population: as for outcome 7
Measure: Median (Full Range); unit: hour
Arm/Group | Japanese Cohort 1: TAK-831 100 mg | Japanese Cohort 1: TAK-831 300 mg | Japanese Cohort 2: TAK-831 300 mg | Japanese Cohort 4: TAK-831 600 mg | Japanese Cohort 5: TAK-831 50 mg | Chinese Cohort 3: TAK-831 600 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
hour
  Day 1 | 0.5000 [0.500 to 0.500] | 0.5000 [0.500 to 1.00] | 2.000 [1.50 to 4.00] | 1.750 [1.50 to 4.00] | 0.5000 [0.500 to 1.50] | 1.500 [1.50 to 2.00]
  Day 17 | NA [NA to NA] — Tmax for Cohort 1 was not planned to analyzed on Day 17. | NA [NA to NA] — Tmax for Cohort 1 was not planned to analyzed on Day 17. | 1.750 [1.00 to 4.000] | 2.000 [1.00 to 4.00] | 0.5000 [0.500 to 2.00] | 2.000 [1.50 to 2.00]

9. Secondary Outcome: AUClast: Area Under the Plasma Concentration-time Curve (AUC) From Time 0 to Time of the Last Quantifiable Concentration for TAK-831
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter(h*ng/mL)
Arm/Group | Japanese Cohort 1: TAK-831 100 mg | Japanese Cohort 1: TAK-831 300 mg | Japanese Cohort 2: TAK-831 300 mg | Japanese Cohort 4: TAK-831 600 mg | Japanese Cohort 5: TAK-831 50 mg | Chinese Cohort 3: TAK-831 600 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
hour*nanogram per milliliter(h*ng/mL) | 1553 (11.8) | 3630 (11.9) | 3700 (32.2) | 6477 (26.2) | 847.4 (21.5) | 5504 (22.3)

10. Secondary Outcome: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-831
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Japanese Cohort 1: TAK-831 100 mg | Japanese Cohort 1: TAK-831 300 mg | Japanese Cohort 2: TAK-831 300 mg | Japanese Cohort 4: TAK-831 600 mg | Japanese Cohort 5: TAK-831 50 mg | Chinese Cohort 3: TAK-831 600 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
h*ng/mL | 1581 (11.7) | 3653 (12.2) | 3730 (31.9) | 6518 (26.2) | 923.6 (22.1) | 5530 (22.3)

11. Secondary Outcome: Cohorts 2 to 5, AUCtau: Area Under the Plasma Concentration-time Curve From Time 0 to [Time] Over the Dosing Interval for TAK-831
Time Frame: Day 1: pre-dose and at 0.25, 0.5, 1, 1.5, 2, 4, 8, 12, 24, 36, 48 and 72 hours post-dose and Day 17: pre-dose and at 0.25, 0.5, 1, 1.5, 2, 4, 8, 12, and 24 hours post-dose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Japanese Cohort 2: TAK-831 300 mg | Japanese Cohort 4: TAK-831 600 mg | Japanese Cohort 5: TAK-831 50 mg | Chinese Cohort 3: TAK-831 600 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
h*ng/mL
  Day 1 | 3576 (30.6) | 6211 (26.8) | 794.5 (22.2) | 5340 (22.3)
  Day 17 | 2738 (31.1) | 8237 (28.4) | 983.0 (22.3) | 5839 (21.6)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of study drug up to Day 23 in Cohort 1 and up to Day 31 in Cohorts 2 to 5
Arm/Group | Japanese Cohort 1: Placebo | Japanese Cohort 1: TAK-831 100 mg | Japanese Cohort 1: TAK-831 300 mg | Japanese Cohort 2, 4 and 5: Pooled Placebo | Japanese Cohort 2: TAK-831 300 mg | Japanese Cohort 4: TAK-831 600 mg | Japanese Cohort 5: TAK-831 50 mg | Chinese Cohort 3: Placebo | Chinese Cohort 3: TAK-831 600 mg
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/2 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/2 | 0/6
Other Adverse Events (participants affected / at risk) | 0/4 | 2/6 | 0/6 | 4/6 | 4/6 | 1/6 | 2/6 | 1/2 | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Japanese Cohort 1: Placebo (N=4) | Japanese Cohort 1: TAK-831 100 mg (N=6) | Japanese Cohort 1: TAK-831 300 mg (N=6) | Japanese Cohort 2, 4 and 5: Pooled Placebo (N=6) | Japanese Cohort 2: TAK-831 300 mg (N=6) | Japanese Cohort 4: TAK-831 600 mg (N=6) | Japanese Cohort 5: TAK-831 50 mg (N=6) | Chinese Cohort 3: Placebo (N=2) | Chinese Cohort 3: TAK-831 600 mg (N=6)
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Protein urine present (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Procedural headache (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Vascular procedure complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0
Blood pressure systolic increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Red blood cells urine positive (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
White blood cells urine positive (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, the PI may publish results of the study following the publication of results by the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2019-02-26): https://cdn.clinicaltrials.gov/large-docs/84/NCT03687684/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-27): https://cdn.clinicaltrials.gov/large-docs/84/NCT03687684/SAP_001.pdf